CLINICAL TRIAL: NCT06854575
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Nutraceutical Supplement With Standardized Botanicals in Aging Males With Thinning Hair
Brief Title: A Safety and Efficacy Study of a Nutraceutical in Aging Males With Thinning Hair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Business Decision
Sponsor: Nutraceutical Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NW-MSS-01
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Hair Thinning
MeSH Terms: conditions — Alopecia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Dietary Supplement
  Interventions: Dietary Supplement: Dietary Supplement
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — Oral dietary supplement
  Arms: Active
Other: Placebo — Placebo pill
  Arms: Placebo

SUMMARY:
A study to assess the safety and efficacy of a dietary supplement when used over the course of 9 months by men with self-perceived hair thinning.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled clinical trial is being conducted to assess the safety and efficacy of a dietary supplement with standardized botanicals compared to a placebo when used over the course of 9 months by men with self-perceived hair thinning.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 40 to 65 years of age.
2. In good general health (physical, mental, and social well-being, not merely the absence of disease/infirmity), according to subject self-report.
3. Having Fitzpatrick skin type I-IV.
4. Having overall hair thinning (diffuse thinning of the top of the crown or at temples and/or widening part or receding hair line) confirmed by the study dermatologist at baseline (grade III, IIIa, III vertex, IV, or IVa on the Hamilton-Norwood scale).
5. With self-perceived thinning hair on the scalp.
6. Willing to participate in the Hair Pull Test, in which a trained practitioner will grasp a 4-6mm bundle of hair near the scalp and firmly tug the hair.
7. Having a regular mild, non-medicated shampoo and conditioner (if used) and willing to bring the product(s) in to the first clinic visit for documentation and to continue using the product(s) for the duration of the study.
8. Willing to continue using regularly used hair styling products (mousse, hairspray) if used, and not start using any new hair products for the duration of the study.
9. Willing to maintain the same hair length, hairstyle, and coloring practices for the duration of the study. Those with color-treated hair must have the color treatment performed at the same time interval prior to each visit.
10. Willing to maintain current diet (eg, amount, type, and frequency of food and drink consumed).
11. Willing to not wear hats, scarves, or other head coverings on your head during each study visit.
12. Willing to refrain from using any topical hair products or treatments on the hair that could affect hair properties (eg, heat treatments, hair relaxers, permanent wave, medicated shampoo, etc) for the duration of the study except for the test material and regular shampoo and conditioner (if used) and styling products.
13. Willing to refrain from hair extensions, tight braids, or hair weaves for the duration of the study.
14. Willing to refrain from taking any vitamins, minerals, or herbal supplements with claims related to hair growth or benefits during the study, and to not start taking any new vitamins, minerals, or supplements of any kind during the study.
15. Willing to avoid using prescription or over-the-counter (OTC) products designed to or claiming to significantly impact hair loss and/or hair growth for the duration of the study.
16. Willing to complete a questionnaire regarding sexual experiences (commonly used in clinical trials to assess sexual functioning).
17. Willing to provide written informed consent and able to read, speak, write, and understand English.
18. Willing to sign a photography release.
19. Willing to cooperate and participate by following study requirements for the duration of the study and to report any changes in health status or medications, AE symptoms, or reactions immediately.

Exclusion Criteria:

1. Having a pregnant partner or a partner that is planning to become pregnant during the study.
2. Having a known allergy to any ingredients in the test products.
3. Having a history of skin cancer within the past 5 years.
4. Having hair extensions, hair weave, tight braids, crew cut, or very short hair (less than 1.5 inches in length).
5. Having started any new vitamin, mineral, or herbal supplement within 30 days prior to baseline.
6. Smokers with usage >20 cigarettes/day.
7. Who have been diagnosed with hair loss disorders such as alopecia areata, scarring alopecia, traction alopecia, chemical alopecia, trichotillomania or trichorrhexis nodosa, or suffering from moderate to severe hair loss disorder (grade V-VII on the Hamilton-Norwood scale) confirmed by the investigator.
8. Having hair loss due to disease, injury, or medical therapy.
9. Who have a history of hair transplants or surgical procedures to the head that may have impacted skin anatomy (eg, flaps, grafts, plugs).
10. Who have very brittle or severely damaged hair from causes including chemical treatments and excessive tension on the hair (from, eg, tight ponytails or hair extensions).
11. Having a history of persistent burning, itching, or stinging of the scalp.
12. Having clinically active bacterial, fungal, or viral skin infections or those who have a history of skin infections, according to subject self-report.
13. Who are currently using, planning to use, or have used laser/light therapy (such as HairMax, iRestore), microneedling or scalp micropigmentation, or used any prescription or over-the-counter (OTC) products designed to or claiming to significantly impact hair loss and/or hair growth (eg, minoxidil, Rogaine, finasteride, Propecia, Nioxin shampoo, or oral supplements (such as Biotin >500mcg or Nutrafol)) within 6 months of study start.
14. Having not used any prescription or over-the-counter (OTC) products designed to or claiming to significantly impact hair loss and/or hair growth (eg, minoxidil, Rogaine, finasteride, Propecia, Nioxin shampoo, or oral supplements (such as Biotin >500mcg or Nutrafol) for at least 6 months prior to baseline, and willing to avoid all such products for the duration of the study.
15. Who are currently using, planning to use, or have used anabolic-androgenic steroids (testosterones) or anti-androgen medication (such as spironolactone, flutamide, cyproterone acetate, cimetidine) other than oral contraceptives; platelet-rich plasma (PRP) injections; or tamoxifen within 3 months of study start. (Men currently undergoing hormone/testosterone replacement therapy [TRT] can be eligible for the study if they have maintained a stable dose for at least 6 months prior to enrollment and stay on the same dose throughout the study.)
16. Having started blood pressure medications or aldactone within 3 months of enrollment.
17. Having a health condition and/or pre-existing or dormant dermatologic disease on the scalp (eg, excessive dandruff, psoriasis, eczema, seborrheic dermatitis, severe excoriations) that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
18. Having observable sunburn, suntan, scars, nevi, tattoos, or other dermal conditions on the scalp that might influence the test results in the opinion of the Investigator or designee.
19. Having a history of immunosuppression/immune deficiency disorders (including HIV infection, AIDS, multiple sclerosis, Crohn's disease, rheumatoid arthritis), organ transplant (heart, kidney, etc), or currently using oral or systemic immunosuppressive medications and biologics (eg, azathioprine, belimumab, Cimzia, Cosentyx, cyclophosphamide, cyclosporine, Enbrel, Humira, Imuran, Kineret, mycophenolate mofetil, methotrexate, Orencia, prednisone, Remicade, Rituxan, Siliq, Simponi, Stelara, Taltz) and/or undergoing radiation or chemotherapy as determined by study documentation.
20. Currently using or having regularly used corticosteroids (systemic or topical, not nasal or ocular) within the past 4 weeks (including but not limited to betamethasone, clobetasol, desoximetasone, diflorasone, fluocinonide, halcinonide, and halobetasol).
21. Having a disease such as asthma, diabetes, epilepsy, hypertension, hyperthyroidism, or hypothyroidism that is not controlled by diet or medication. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
22. Having started a long-term medication within the last 2 months.
23. Having any planned surgeries or invasive medical procedures during the study. Noninvasive medical procedures or surgeries will be reviewed for their impact on the study outcome and acceptability by the Investigator or designee.
24. Currently participating in any other clinical trial at SGS or another research facility or doctor's office.
25. Having a history of unstable, not controlled, or chronic depression or bipolar disease or any other disorder that may impact the participation in the study, according to subject self-report.
26. Having a self-reported history of recent blood work indicating iron deficiency, bleeding disorders, or platelet dysfunction syndrome or currently receiving anticoagulant therapy.
27. Having participated in any clinical trial involving the scalp and/or hair within 2 weeks before study enrollment at SGS or another research facility or doctor's office.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population will comprise only of adult men.
Enrollment: 155 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Hair Growth Global Improvement Scale rating at 6 months | 6 months
  Blinded Investigator mean Hair Growth Global Improvement Scale rating at 6 months for treatment group as compared to placebo

SECONDARY OUTCOMES:
Investigator Hair Quality Global Improvement Scale at 6 month | 6 months
  Blinded Investigator Hair Quality Global Improvement Scale mean score at 6 months for treatment group as compared to placebo

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - SGS Phoenix Research Center, Phoenix, Arizona
  - SGS Elizabeth Research Center, Elizabeth, New Jersey
  - SGS Dallas Research Center, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No